CLINICAL TRIAL: NCT05429606
Title: Effect of Different Water-based and Gel-based Conductive Media on the Efficacy of Electric Pulp Tester
Brief Title: Effect of Different Conductive Media on the Efficacy of Electric Pulp Tester
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, nosheen sarwar, Principle Investigator, Pakistan Institute of Medical Sciences
Other Study IDs: SOD/ERB/2022/06
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Healthy Maxillary Central Incisors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: Fluoride gel: The fluoride gel used as conductive media for electric pulp tester in this group
- Group 2:Electrode gel: In Group 2 electrode gel applied as conductive media for electric pulp test.
- Group 3: chlorohexidine gluconate gel: chlorohexidine gluconate gel used as conductive media for electric pulp tester in group 3.
- Group 4:Colgate gel toothpaste: Colgate gel toothpaste gel used as conductive media for electric pulp tester in group 4.
- Group 5:Dentonic Ultrawhitening gel: Dentonic Ultrawhitening gel used as a conductive media in Group 5.

SUMMARY:
Dental pulp tests are investigations that offer valuable diagnostic and treatment planning information to the dental clinician. EPT is a sensibility test that can be easily performed in clinical practice. Current study is to find the best conducting substance among readily available water-based gels and gel-based tooth pastes to evaluate the efficacy of electric pulp tester.

DETAILED DESCRIPTION:
The study will be performed on dental students with written informed constant. The sample size of study is 100. There will two main groups of conductor materials used in the study: water-based gels (fluoride gel, electrode gel and chlorohexidine gluconate) and gel-based toothpastes (Colgate and Dentonic Ultrawhitening gel). All groups will be randomly applied to the same patient at a single visit. Two measurements will be recorded for each material and the average value of the two measurements will used. Then, the measurements will record, and a comparison will be made between different conductors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy fully erupted teeth maxillary central incisors.
* Study subjects above 18 years.
* No systemic diseases and pregnancy

Exclusion Criteria:

* Carious, decayed and periodontally affected teeth.
* Taking anti-inflammatory drugs from last 2 weeks.
* Taking cortisone for the last 6 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study subjects are dental students of School of dentistry Islamabad
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of electric pulp tester | immediately after procedure
  To measure the efficacy of electric pulp tester with different conductive media.

SECONDARY OUTCOMES:
Effect of gender on efficacy of electric pulp tester. | immediately after procedure
  To measure the efficacy based of gender in study subjects

CONTACTS AND LOCATIONS:
Overall Officials: nosheen sarwar, BDS, Principal Investigator — School of dentistry PIMS
Locations (1):
- School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No